CLINICAL TRIAL: NCT03542812
Title: Pharmacokinetics of L-citrulline in Infants at High Risk of Developing Pulmonary Hypertension Associated With Bronchopulmonary Dysplasia
Brief Title: L-citrulline and Pulmonary Hypertension Associated With Bronchopulmonary Dysplasia
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study stopped enrollment prior to the initially projected 18 subjects per phase due to lack of funding to continue to recertify the drug and because an adequate number of subjects were enrolled for each phase to analyze pharmacokinetics.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Candice Fike, Principal Investigator, University of Utah
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 97293
Record Dates: First submitted 2018-05-02; First posted 2018-05-31 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-05

CONDITIONS: Infant,Premature; Bronchopulmonary Dysplasia; Pulmonary Hypertension
Keywords: L-citrulline; Nitric oxide
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia; Hypertension, Pulmonary | interventions — Citrulline

STUDY DESIGN:
Intervention Model Description: Single dose pharmacokinetic studies using population PKs Steady-state pharmacokinetic studies using population PKs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single-dose (Experimental): Participants will be enrolled into the two groups, Group 1 (which will consist of 10 participants) and Group 2 (which will consist of 8 participants) in an alternating basis. Both Group 1 and Group 2 participants will receive a single, 150 mg/kg dose of oral L-citrulline. Population PKs will be done for both groups, at up to 3 time points.
  Multiple interim time points and following completion of enrollment into Groups 1 and 2, data analysis will be done and results reviewed by the data safety monitoring board (DSMB). After the DSMB review is complete, enrollment into Group 3 will begin.
  Interventions: Drug: L-Citrulline
- Steady-state (Experimental): To evaluate the tolerability and ability to achieve target trough L-citrulline levels of 100-150 µM, an additional group of 18 infants (group 3) will be given oral L-citrulline doses at intervals over a total of 72 hours. If the participant is not nipple feeding, the dose will be delivered via the participant's indwelling gavage feeding tube. The dose and interval of L-citrulline will be based on results from the studies that assess pharmacokinetic parameters using a maximum daily dose of 3 g/kg/d. Blood draws for PKs will be done at baseline and prior to last dose of L-citrulline. Urine will be collected to measure nitric oxide metabolites.
  Interventions: Drug: L-Citrulline

INTERVENTIONS:
Drug: L-Citrulline — The L-citrulline will be procured in powder form and will be solubilized in sterile water to achieve a concentration of 50 mg/ml. Therefore, 3 ml/kg of the solubilized L-citrulline (50 mg/ml) will be administered per dose for the single-dose groups and the dose administered to the steady-state group will be determined from results from the single-dose studies.

SUMMARY:
Bronchopulmonary dysplasia (BPD) is a chronic lung disease that affects up to 35% of very low birth weight infants (VLBW < 1500 g). Based on the current numbers of VLBW infants born annually in the U.S., between 5,000-10,000 neonates will develop BPD each year. It is estimated that 8-42% of infants with BPD will develop pulmonary hypertension (PH). Moreover, it has been known since the 1980's that echocardiographic evidence of PH in infants with BPD is associated with up to 40% mortality.

Treatment options to ameliorate PH in infants with BPD (BPD-PH) are limited. There have been no randomized clinical trials of any therapy in infants with BPD-PH. The standard care for the management of BPD-PH is to attempt to resolve the underlying lung disorder and the judicious use of oxygen as a potent pulmonary vasodilator. Using this management approach, which has not changed since the 1980's, the survival rates for infants with BPD-PH in the 2000's has been reported to be 64% at 6 months and 53% at 2 years after diagnosis of PH. The lack of improvement in outcomes for the past 3 decades has led to the widespread agreement that novel and effective therapies are desperately needed for infants with BPD-PH.

The goal is to develop oral L-citrulline clinically for the treatment of pediatric pulmonary hypertension associated with bronchopulmonary dysplasia (BPD-PH); before pursuing a large scale treatment trial, pharmacokinetic (PK) dose-finding, tolerability studies in patients at high risk of developing BPD-PH are warranted.

The hypothesis is that oral L-citrulline will be well tolerated, without significant adverse effects in infants at high risk of developing pulmonary hypertension (PH) associated with BPD. The investigators propose to first characterize the PK profile of oral L-citrulline in order to define an appropriate dose range and treatment interval for infants at high risk of developing BPD-PH. Then using the doses and intervals generated by the PK profile, with a maximum dose of 3 g/kg/d, the investigators propose to evaluate the tolerability and ability to achieve the target study drug level (100-150 micromolar) in babies treated for 72 hours with oral L-citrulline. These studies will provide the data needed to design a full-scale randomized multi-center trial to evaluate the efficacy of oral L-citrulline therapy to ameliorate BPD-PH in human infants, a patient population that has a desperate need of new therapies.

ELIGIBILITY:
Inclusion Criteria:

Infants born prematurely at < or = 28 weeks gestation requiring invasive (mechanical ventilation) or non-invasive positive pressure support (nasal continuous positive airway pressure, high flow nasal cannula >1 lpm) and FiO2 of at least 0.30 at 32 +/- 1 weeks postmenstrual age

2.Tolerating at least one-half of full volume oral/gavage tube feedings (using 120 ml/kg/d as full volume oral/gavage tube feedings)

3.The continuous need for some form of respiratory support (supplemental oxygen, flow) for the prior 14 days

4.Hemoglobin > 10 mg/dL

Exclusion Criteria:

1. Known major fetal anomaly or chromosomal aneuploidy
2. Clinical evidence of congenital heart disease (except patent ductus arteriosus (PDA), atrial septal defect (ASD), or ventricular septal defect (VSD)
3. Urine output < 1 ml/kg/hr
4. History of or known to have liver failure
5. History of or known to have necrotizing enterocolitis
6. History of or known to have significant feeding intolerance beyond the first week of life
7. Presence of any acute illness defined by fever >100.4 F, vomiting, or diarrhea
8. Hemoglobin < 10 mg/dL
9. Neonatal Intensive Care Unit (NICU) cases determined to be futile (anticipated death prior to hospital discharge)
10. Multiple births

Ages: 14 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Candice Fike, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fike CD, Avachat C, Birnbaum AK, Aschner JL, Sherwin CM. Pharmacokinetics of L-Citrulline in Neonates at Risk of Developing Bronchopulmonary Dysplasia-Associated Pulmonary Hypertension. Paediatr Drugs. 2023 Jan;25(1):87-96. doi: 10.1007/s40272-022-00542-x. Epub 2022 Oct 31. PMID 36316628
- [Result] Fike CD, Aschner JL, Avachat C, Birnbaum AK, Sherwin CMT. Multi-dose enteral L-citrulline administration in premature infants at risk of developing pulmonary hypertension associated with bronchopulmonary dysplasia. J Perinatol. 2024 Feb;44(2):280-287. doi: 10.1038/s41372-023-01809-y. Epub 2023 Oct 31. PMID 37907796
- [Derived] Aschner J, Avachat C, Birnbaum A, Sherwin C, Fike C. Multi-dose enteral L-citrulline administration in premature infants at risk of developing pulmonary hypertension associated with bronchopulmonary dysplasia. Res Sq [Preprint]. 2023 Jun 9:rs.3.rs-3006963. doi: 10.21203/rs.3.rs-3006963/v1. PMID 37333204

RESULTS

PARTICIPANT FLOW:
Groups:
- Single-dose: Participants will be enrolled into the two groups, Group 1 (which will consist of 10 participants) and Group 2 (which will consist of 8 participants) in an alternating basis. Both Group 1 and Group 2 participants will receive a single, 150 mg/kg dose of oral L-citrulline. Population PKs will be done for both groups, at up to 3 time points.
  Multiple interim time points and following completion of enrollment into Groups 1 and 2, data analysis will be done and results reviewed by the data safety monitoring board (DSMB). After the DSMB review is complete, enrollment into Group 3 will begin.
  L-Citrulline: The L-citrulline will be procured in powder form and will be solubilized in sterile water to achieve a concentration of 50 mg/ml. Therefore, 3 ml/kg of the solubilized L-citrulline (50 mg/ml) will be administered per dose for the single-dose groups and the dose administered to the steady-state group will be determined from results from the single-dose studies.
Period: Overall Study
Arm/Group | Single-dose | Steady-state
Started | 10 | 6
Completed | 10 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single-dose | Steady-state | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 6 | 16
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: Post-menstrual age in weeks at study] | 31.4 [31.4 to 32.4] | 32.0 [31.1 to 33.0] | 31.7 [31.1 to 33.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 8 | 4 | 12
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 4 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Plasma L-citrulline Levels Following Administration of a Single Dose of L-citrulline- Arm 1
Description: Plasma L-citrulline levels will be measured using population pharmacokinetics (PK) before and at intervals following administration of a single dose of oral L-citrulline and used to generate a population pharmacokinetic model in patients at high risk of developing BPD-PH. This arm will be split into two groups of 5 subjects each. Group 1 will have PKs done at baseline (24-48 hours prior to first dose), 1 hour (+/- 10 minutes) after dose given and 2.5 hours (+/- 10 minutes) after dose given. Group 2 will have PKs done at baseline (24-48 hours prior to first dose), 15 minutes (+/- 10 minutes) after dose given and 3 hours (+/- 10 minutes) after dose given.
Time Frame: Group 1- Baseline, 1 hr post-study drug dose, and 2.5 hours post-study drug dose, Group 2- Baseline, 15 minutes post-study drug dose and 3 hours post-study drug dose
Population: All babies in this arm had a baseline level PK. Group 1 (5 subjects) had a PK done at 1 hour (+/- 10 minutes) after dose given and 2.5 hours (+/- 10 minutes) after dose given. Group 2 (5 subjects) had a PK done at 15 minutes (+/- 10 minutes) after dose given and 3 hours (+/- 10 minutes) after dose given.
Measure: Median (Full Range); unit: micromol/L
Groups:
- Single-dose Group, Baseline L-citrulline Levels: Blood was sampled from all subjects 24-48 hours prior to the first study drug dose of L-citrulline and measured for baseline L-citrulline levels.
- Single-dose Group, L-citrulline Level 15 Min After Study Drug: Blood was sampled from 5 subjects at 15 min after study drug L-citrulline was given +/- 10 minutes.
- Single-dose Group, L-citrulline Level at 1 Hour After Study Drug: Blood was sampled from 5 subjects at 1 hour after study drug L-citrulline was given +/- 10 minutes.
- Single-dose Group, L-citrulline Level at 2.5 Hours After Study Drug: Blood was sampled from 5 subjects at 2.5 hours after study drug L-citrulline was given +/- 10 minutes.
- Single-dose Group, L-citrulline Level at 3 Hours After Study Drug: Blood was sampled from 5 subjects at 3 hours after study drug L-citrulline was given +/- 10 minutes.
Arm/Group | Single-dose Group, Baseline L-citrulline Levels | Single-dose Group, L-citrulline Level 15 Min After Study Drug | Single-dose Group, L-citrulline Level at 1 Hour After Study Drug | Single-dose Group, L-citrulline Level at 2.5 Hours After Study Drug | Single-dose Group, L-citrulline Level at 3 Hours After Study Drug
Number analyzed (Participants) | 10 | 5 | 5 | 5 | 5
micromol/L | 31 [9 to 36] | 470 [340 to 554] | 651 [388 to 799] | 232 [189 to 507] | 197 [97 to 224]

2. Primary Outcome: Evaluate L-citrulline Plasma Levels at Baseline and Prior to the Last Dose of Study Drug Dose (Dose #12)- Arm 2
Description: Evaluate the ability to achieve the target trough L-citrulline plasma level of approx.50-80 µM in patients at high risk of developing BPD-PH treated for 72 hours with oral L-citrulline by measuring baseline L-citrulline levels and L-citrulline plasma levels drawn prior to last dose of L-citrulline study drug. Study drug is given orally every 6 hours over 72 hours for a total of 12 doses. A PK will be done on all subjects at baseline (10 minutes to 6 hours prior to first dose) and again 10-30 minutes prior to last dose. If all 12 doses of study drug are given, this will be at approximately 65.5 hours after the first study drug dose is given.
Time Frame: 10 min to 1 hour prior to first study drug dose and 10-30 minutes prior to last dose (approx 65.5 hours after the first dose given).
Population: All subjects had a baseline PK and trough PK done prior to 12th dose (approx 65.5 hours after first dose of study drug)
Measure: Median (Inter-Quartile Range); unit: micromol/L
Groups:
- Steady-state Group, Baseline L-citrulline Plasma Concentrations: Blood samples were obtained from all subjects 24-48 hours prior to first study drug L-Citrulline dose
- Steady-state Group, Trough Level Prior to Last Study Drug L-citrulline Dose: Blood samples were obtained prior to last study drug L-citrulline dose (dose #12) and L-citrulline levels were measured.
Arm/Group | Steady-state Group, Baseline L-citrulline Plasma Concentrations | Steady-state Group, Trough Level Prior to Last Study Drug L-citrulline Dose
Number analyzed (Participants) | 6 | 6
micromol/L | 37.5 [20 to 45] | 38 [30.5 to 53]

3. Primary Outcome: Number of Participants With Feedings Being Stopped Following L-citrulline Administration
Description: The safety outcome of the tolerability of L-citrulline will be measured by whether a subject has feedings held within 48 hours of receiving oral L-citrulline administration for reasons not attributable to underlying condition. For the stead state arm, feeding tolerance was monitored during the 72 hour period in which study was given and then for another 48 hours after the last study drug was given.
Time Frame: 48 hours after last study drug dose
Measure: Count of Participants; unit: Participants
Groups:
- Single-dose: All subjects were monitored for 48 hours after single dose of 150 mg/kg L-citrulline given orally to evaluate evidence of intolerance by having feedings stopped.
- Steady-state: All subjects were monitored during the 72 hours of receiving study drug and for 48 hours after the last dose of study drug L-citrulline given orally to evaluate evidence of intolerance by having feedings stopped.
Arm/Group | Single-dose | Steady-state
Number analyzed (Participants) | 10 | 6
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Hypotension Developing Following L-citrulline Administration
Description: The safety outcome of tolerability of L-citrulline will be measured by whether a subject develops a decrease in blood pressure more than 25% below baseline within 12 hours of receiving a dose of oral L-citrulline for reasons not attributable to underlying condition
Time Frame: 12 hours after last study drug dose
Measure: Count of Participants; unit: Participants
Groups:
- Single-dose: All subjects were monitored for 48 hours after single dose of 150 mg/kg L-citrulline given orally to evaluate for evidence of hypotension by measuring blood pressures every 12 hours.
- Steady-state: All subjects were monitored during the 72-hour administration period and for 48 hours after last dose of study drug L-citrulline given orally to evaluate for evidence of hypotension by measuring blood pressures every 12 hours.
Arm/Group | Single-dose | Steady-state
Number analyzed (Participants) | 10 | 6
Participants | 0 | 1

5. Secondary Outcome: Urinary Nitrite and Nitrate Levels Will be Measured in Subjects Enrolled Into the Steady State (Second Arm) of the Study.
Description: Urine samples will be obtained to assess baseline levels of nitric oxide metabolites (nitrite/nitrate) in the urine within 24 hours prior to first dose and again 4-8 hours after the last dose of study drug given. The purpose is to assess whether there is an increase in levels of nitric oxide metabolites in the urine in response to 72 hours of L-citrulline dosing. Urine samples are only being obtained in infants enrolled in the steady state (second arm) of the study.
Time Frame: Baseline (within 24 hours prior to first study drug dose) and 4-8 hours after last study drug dose given (approximately 70 to 78 hours after first study drug dose)
Population: Only subjects in the steady state arm (second arm) of the study had urine analyzed. 1 subject only had post-study urine available for analysis so this subject was not included in the overall analysis.
Measure: Median (Inter-Quartile Range); unit: micromol/g Cr
Groups:
- Steady-state Group, Baseline NOx/Cr Levels: Urine was collected prior the first dose of oral L-citrulline to measure the NOx/Cr levels.
- Steady-state Group; NOx/Cr Levels in Urine After Last Study Drug Dose: Urine was collected 6-7 hours after last dose of L-Citrulline and the NOx/Cr levels were evaluated.
Arm/Group | Steady-state Group, Baseline NOx/Cr Levels | Steady-state Group; NOx/Cr Levels in Urine After Last Study Drug Dose
Number analyzed (Participants) | 5 | 5
micromol/g Cr | 25.8 [22 to 44] | 36 [27 to 46.6]

ADVERSE EVENTS:
Time Frame: Subjects will be monitored for the duration of study drug receipt and for another 48 hours after last study drug dose given for all AEs with the exception of hypotension, which will be followed for 12 hours after the last study drug dose.
Description: There were two adverse events of special interest: Feeding tolerance and hypotension. All other AEs were only collected if they met the definition of being serious and/or unexpected for the study population and/or related or probably related to the participation in the study.
Arm/Group | Single-dose | Steady-state
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 0/10 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-dose (N=10) | Steady-state (N=6)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) — Mean blood pressure decreased more than 25% of baseline x 1 blood pressure done around dose #3. Infant was asymptomatic and not treated and blood pressure was back to baseline with next measurement 6 hours later. No further low blood pressures.

LIMITATIONS AND CAVEATS:
The study was terminated prior to full enrollment goals of group 3 (steady-state group), therefore there was a small number of subjects for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT03542812/Prot_SAP_000.pdf